CLINICAL TRIAL: NCT07031986
Title: One-lung Ventilation With Double-Lumen Tubes and Bronchial Blockers in Obese Patients Undergoing Lung Resection
Brief Title: Bronchial Blockers vs Double-Lumen Tubes in Obese Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paulo Andrés Cano Jiménez (Other)
Responsible Party: Sponsor-Investigator, Paulo Andrés Cano Jiménez, Principal Investigator, Hospital Son Espases
Organization: Hospital Son Espases (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IB 5484/24 PI
Record Dates: First submitted 2025-06-11; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: One-lung Ventilation
Keywords: one-lung ventilation; lung resection; bronchial blocker; double-lumen tube
MeSH Terms: interventions — One-Lung Ventilation

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to one of two one-lung ventilation groups. The study focuses on intraoperative ventilation during lung resection; therefore, no follow-up is planned. The study concludes for each patient at the end of the surgery.
Who Masked: Participant
Masking Description: Patients do not know which device will be used during their surgery, as is typical in routine clinical practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bronchial Blocker (Experimental): Patients undergoing lung resection who receive one-lung ventilation using a bronchial blocker.
  Interventions: Device: One-Lung Ventilation with Bronchial Blocker
- Double-Lumen Tube (Experimental): Patients undergoing lung resection who receive one-lung ventilation using a double-lumen tube.
  Interventions: Device: One-Lung ventilation with Double-Lumen Tube

INTERVENTIONS:
Device: One-Lung ventilation with Double-Lumen Tube — To achieve the required one-lung ventilation during lung resection, patients will be managed with a double-lumen tube.
  Arms: Double-Lumen Tube
Device: One-Lung Ventilation with Bronchial Blocker — To achieve the required one-lung ventilation during lung resection, patients will be managed with a bronchial blocker.
  Arms: Bronchial Blocker

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of bronchial blockers and double-lumen tubes in achieving one-lung ventilation in obese patients undergoing lung resections. The primary question it aims to answer is:

• Is intraoperative hypoxia significantly different depending on the device used?

Researchers will compare the use of bronchial blockers and double-lumen tubes to assess differences in efficacy and safety.

Participants will not be required to perform any tasks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2
* Diagnostic or clinical suspicion of lung cancer
* Lung resection surgery (lobectomy, segmentectomy or wedge resection) by VATS or thoracotomy, requiring one-lung ventilation.
* Use of bronchial blocker or double-lumen tube for one-lung ventilation.

Exclusion Criteria:

* Patients with evident anatomic alterations, in which double-lumen tubes may be contraindicated.
* Emergency surgeries.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Hypoxia | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  While its definition is somewhat arbitrary, the investigators consider hypoxia as SpO₂ < 90%, while maintaining FiO₂ = 1.0, in accordance to our hospital guidelines.

SECONDARY OUTCOMES:
Lung collapse | Intraoperative
  Assessed by the anaesthesiologist as: Excellent: complete lung collapse, perfect surgical visualization; Good: complete collapse, residual air; Poor: non-achieved collapse or partial collapse that interfered with surgical visualization.
Surgical visualization | Intraoperative
  Assessed by the thoracic surgeon as excellent, good or poor.
Insertion time of the ventilation device | Intraoperative
  Time in minutes from the beginning of ventilation device insertion until correct placement is confirmed.
Repositioning of the ventilation device | Intraoperative
  Number of repositioning attempts of the ventilation device.
Ventilation device change | Intraoperative
  When ventilation cannot be achieved with the device randomly allocated to the patient, conversion to the alternative device must be documented.
Techniques employed in case of hypoxia | Intraoperative
  Record of intraoperative interventions performed in response to hypoxia (defined as SpO₂ < 90% despite FiO₂ = 1.0), including: increase in FiO₂, VENTRAIN ventilation/oxygenation, continuous positive airway pressure (CPAP) to the non-dependent lung, or temporary return to bilateral lung ventilation.
SpO₂ | Preoperative and intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Peripheral oxygen saturation, measured as a percentage.
Ventilation mode | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Type of mechanical ventilation mode applied intraoperatively, categorized as volume-controlled ventilation (VCV), pressure-controlled ventilation (PCV), or pressure-controlled ventilation with volume guarantee (PCV-VG).
Tidal volume (Vt) | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Volume of air delivered to the lungs with each ventilator breath during mechanical ventilation (mL).
Respiratory Rate (Fr) | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Number of ventilator-delivered breaths per minute (bpm) during intraoperative mechanical ventilation.
Peak Airway pressure | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Maximum pressure reached during inspiration in mechanical ventilation, reflecting resistance in the airways (cmH₂O).
Plateau Pressure | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Pressure measured during an inspiratory pause (cmH₂O).
Driving Pressure | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Difference between plateau pressure and positive end-expiratory pressure (cmH₂O).
Fraction of Inspired Oxygen (FiO₂) | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Percentage of oxygen in the gas mixture delivered by the ventilator during mechanical ventilation.
Partial Pressure of Arterial Oxygen (PaO₂) | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Measurement of arterial oxygen tension during mechanical ventilation (mmHg).
Partial Pressure of Arterial Carbon Dioxide (PaCO₂) | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Measurement of arterial carbon dioxide tension (mmHg).
PaO₂/FiO₂ | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Ratio of arterial oxygen partial pressure to the fraction of inspired oxygen.
Hemoglobin | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Arterial blood concentration of hemoglobin, collected intraoperatively as part of blood gas analysis (g/dL).
Hematocrit | Intraoperative (both from anesthetic induction to one-lung ventilation, and during one-lung ventilation)
  Percentage of red blood cells in whole blood, measured intraoperatively as part of arterial blood gas analysis (%).
Intraoperative complications | Intraoperative
  Type of intraoperative complications related to the airway device, including: displacement of the bronchial blocker, tracheobronchial tree rupture, misplacement, trauma to the tracheobronchial tree, need for conversion to thoracotomy, and other complications.
Postoperative recovery complications | First 24 hours after surgery
  Incidence of complications during the immediate postoperative period, including sore throat, aphonia, and other symptoms related to airway instrumentation.

OTHER OUTCOMES:
Sex | Preoperative
  Male or female.
Age | Preoperative
  Age at the time of the procedure (years).
Obesity | Preoperative
  Categorized as: Grade I (BMI: 30-34.9); Grade II (BMI: 35-35.9); Grade III (BMI≥ 40).
Charlson Comorbidity Index | Preoperative
  The Charlson Comorbidity Index (CCI) is a validated scoring system used to predict 10-year mortality by assigning weighted scores to 19 comorbid conditions, based on their severity. The total score reflects both the number and seriousness of comorbid diseases, with higher scores indicating a greater comorbidity burden. Values range from 0 to 33.
Smoker | Preoperative
  Yes or no.
ASA Scale | Preoperative
  The American Society of Anesthesiologists (ASA) Physical Status Classification assesses the preoperative health status of patients undergoing surgery: ASA I: Normal health; ASA II: Mild systemic disease; ASA III: Severe systemic disease; ASA IV: Severe systemic disease that is constant threat to life; ASA V: Moribund, not expected to survive without operation; ASA VI: Declared brain-dead.
Revised Cardiac Risk Index (RCRI) | Preoperative
  The Revised Cardiac Risk Index (RCRI) estimates a patient's risk of perioperative cardiac complications. It is calculated based patient's comorbidities and the type of surgery. A score from 0 to 6 is assigned based on the number of risk factors present.
Airway Assesment | Preoperative
  Assessed by El-Ganzouri Risk Index, which categorizes the risk of a difficult airway (low or high) by taking into account mouth opening, tyromental distance, Mallampati classification, cervical mobility, pronation, weight and difficult intubation history.
Alveolar recruitment maneuvers | Intraoperative
  Yes or no.
Anesthetics | Intraoperative
  Halogenated or intravenous.
Intubation assistance device | Intraoperative
  Laryngoscope or videolaryngoscope.
Laryngoscopy visualization | Intraoperative
  Cormack-Lehane scale: Grade I (complete visualization of vocal chords); Grade II (partial visualization of vocal chords); Grade III (epiglottis visualization, no visualization of vocal chords); Grade IV (no visualization of epiglottis).
Laterality of the blockage | Intraoperative
  Bronchus in which the device is inserted.
Mask ventilation | Intraoperative
  Han Scale: Grade 0: no mask ventilation; Grade 1: Easy mask ventilation; Grade 2: Needs oral airway or adjuvant with or without neuromuscular blocking agents; Grade 3: Difficult - inadequate or unstable or requiring two care providers, with or without neuromuscular blocking agents; Grade 4: Impossible - unable to mask ventilate with or without neuromuscular blocking agents.
Surgery time | Intraoperative
  Total surgical time in minutes, measured from the first incision to the completion of wound closure.
Lung resection | Intraoperative
  Lobectomy, segmentectomy or wedge resection.
Etiology | Intraoperative
  Malignant or benign lung neoplasia.
VATS procedure | Intraoperative
  Yes or no.
Thoracotomy | Intraoperative
  Yes or no.
Patient positioning | Intraoperative
  Lateral, supine or prone position.
DLCO | Preoperative
  Preoperative diffusion capacity of the lung for carbon monoxide (DLCO), expressed as a percentage of the predicted value.
FEV1 | Preoperative
  Preoperative forced expiratory volume in one second (FEV1), reported as a percentage of the predicted value.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Andrés Cano, MD, Principal Investigator — Hospital Son Espases
Locations (1):
- Hospital Son Espases, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided